CLINICAL TRIAL: NCT05995483
Title: Kendi Kendine Meme Muayenesi Ile İlgili Anımsatıcı Bildirimlerin Meme Kanseri Korkusu ve Sağlık İnançları Üzerine Etkisi/The Effect of Reminder Notifications About Breast Self-Exam on Fear of Breast Cancer and Health Beliefs
Brief Title: Experimental Study With Pretest/Posttest Groups Which the Intervention Group Have the System Which Sends Reminder Notifications Directing Them to the Website Containing BSE Training Along With the Illustrations Created for the Practice Prepared by the Researcher on the Determined Ideal Day
Acronym: BreastSelfExam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ETK00-2022-0030
Record Dates: First submitted 2023-07-18; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Breast Self-Examination; Breast Cancer; Nursing Caries; Cancer; Awakening Early
Keywords: Awareness; Early Diagnosis; Prevent Surgery; Breast Self-Examination
MeSH Terms: conditions — Breast Self-Examination; Breast Neoplasms; Neoplasms; Sleep Initiation and Maintenance Disorders; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Have access to web based BSE training and notifications (Experimental): Have the System Which Sends Reminder Notifications Directing Them to the Website Containing BSE Training Along With the Illustrations Created for the Practice Prepared by the Researcher on the Determined Ideal Day.
  Interventions: Other: Early Diagnosis on BSE
- Has no intervention during the study (No Intervention): Only has an powerpoint training og BSE, not knowing about the web base system

INTERVENTIONS:
Other: Early Diagnosis on BSE — the System Which Sends Reminder Notifications Directing Them to the Website Containing BSE Training Along With the Illustrations Created for the Practice Prepared by the Researcher on the Determined Ideal Day.
  Arms: Have access to web based BSE training and notifications

SUMMARY:
H0: Among the intervention and control groups of reminder notifications relating to self-examination

H01: Average breast cancer fear score and H02: There is no difference in the average score of breast cancer health beliefs.

H1: Among the intervention and control groups of reminder notifications relating to self-examination

H11: Average breast cancer fear score H12: Breast cancer is different in terms of average score of health beliefs

DETAILED DESCRIPTION:
Newly Enrolled Students in the Nursing Programs at Girne American University and Eastern Mediterranean University Will Participate in This Study as an Experimental Study With a Pretest/Posttest Control Group. The Students Will Receive the Same Training. Contrary to the Control Group, the Intervention Group Will Have the System Which Will Send Reminder Notifications (Via the Web Base) Directing Them to the Website Containing BSE Training, Along With the Vector Illustration to be Created for the Concurrent Practice Prepared by the Researcher on the Determined Ideal Day. Users Will Receive a Notification Twice Via the Website and Email That Includes Re-examination Seven Days Following the End of Their Period. Depending on the Permission They Grant to Their Phones, Users Will be Able to Access the BSE Training Materials on the Website by Clicking on the General Reminder Notification or the Router, Using Their Browsers, and Logging in to Their Accounts. The Data on the Frequency of BSE With the "Breast Cancer Fear Scale" and "Champion's Health Belief Model Scale" Will be Collected From the Users at the End of the Three-month Period of Using the Website, Which Will be Developed in Order to Raise the Chances of Early Diagnosis by Encouraging BSE.

ELIGIBILITY:
Inclusion Criteria:

* Who is over 18 years old,
* Eastern Mediterranean University and Girne American University, newly enrolled female students in the Nursing Department of the Faculty of Health Sciences

Exclusion Criteria:

* People who do not meet the criteria

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The research is planned to do on female nursing students
Enrollment: 76 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-09-04 (Estimated); Study Completion 2023-09-04 (Estimated)

PRIMARY OUTCOMES:
Change in the health belief scores on 'Champion Health Belief Model Scale' and 'Breast Cancer Fear Scale' related web based BSE examination notifications in 3 months. | 3 months
  Measuring the health belief on breast cancer early diagnosis and awareness with web based bse training and notifications using 'Champion Health Belief Model Scale' and 'Breast Cancer Fear Scale'.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University & Girne American University, Kyrenia, Cyprus

IPD SHARING:
Plan to Share IPD: Yes